CLINICAL TRIAL: NCT01665794
Title: Multicenter, Open-label, Single-arm, Phase 1b/2 Study of the Safety and Efficacy of Combination Treatment With Pomalidomide, Dexamethasone, and Carfilzomib (PdC) in Subjects With Relapsed and Relapsed/Refractory Multiple Myeloma
Brief Title: Carfilzomib, Pomalidomide, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12-1088; NCI-2012-01168 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; carfilzomib; Dexamethasone; Calcium Dobesilate; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- PdC Group (Experimental): Patients receive carfilzomib, pomalidomide, and dexamethasone at indicated doses and schedule every 28 days. Patients may continue to receive treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pomalidomide; Drug: Carfilzomib; Drug: dexamethasone
- PdC + Dara Group (Experimental): Patients receive carfilzomib, pomalidomide, dexamethasone, and daratumumab at indicated doses and schedule every 28 days. Patients may continue to receive treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pomalidomide; Drug: Carfilzomib; Drug: dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide taken orally at assigned dose.
  Other Names: CC-4047; Pomalyst(R)
Drug: Carfilzomib — Carfilzomib given by intravenous (IV) infusion at assigned dose.
  Other Names: Kyprolis (R); PR-171
Drug: dexamethasone — Dexamethasone taken orally of given by IV infusion.
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: Daratumumab — Daratumumab given by intravenous (IV) infusion at assigned dose.
  Other Names: Daralex
  Arms: PdC + Dara Group

SUMMARY:
The study will investigate the effects of adding carfilzomib to the combination of pomalidomide and dexamethasone in sequential dose escalation cohorts in patients with relapsed or refractory multiple myeloma. This portion of the study is complete.

This study will also investigate the effects of adding daratumumab to the combination of carfilzomib, pomalidomide and dexamethasone.

DETAILED DESCRIPTION:
Patients receive carfilzomib, pomalidomide, and dexamethasone in 28 days treatment cycles. Study treatment continues for as long a their myeloma does not worsen and they do not have unacceptable side effects. After completion of study treatment, patients are followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and relapsed/refractory multiple myeloma requiring systemic therapy
* Failed at least one prior treatment for multiple myeloma (must have received lenalidomide)

  * To be enrolled as second line therapy: Must be refractory to lenalidomide (progression on therapy or within 60 days of lenalidomide dosing)
* Measurable disease, as indicated by one or more of the following:

  * Serum M-protein >= 0.5 g/dL
  * Urine M-protein >= 200 mg/24 hours
  * If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative immunoglobulin levels are acceptable
  * Involved serum free light chains ≥ 10 mg/dL (free light change ratio must be abnormal)
* Aged 18 years or older
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate Liver Function

  * Bilirubin < 1.5 times the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) < 2.5 times ULN
  * Alanine aminotransferase (ALT) < 2.5 times ULN
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 8 g/dL
* Platelet count >= 75 x 10^9/L (should be independent of platelet transfusions for at least 2 weeks)
* Calculated or measured creatinine clearance of >= 30 mL/minute
* Written informed consent
* Negative pregnancy test (for women of childbearing potential) within 10-14 days of starting study treatment and again within 24 hours of first pomalidomide dose
* Must agree to practice abstinence or use two acceptable methods of birth control
* Men must agree to use latex condom during sexual contact with women of childbearing potential (even if post vasectomy)
* Must agree to adhere to all study requirements, visit schedule, outpatient treatment, required concomitant medications, and laboratory monitoring
* Must register to mandatory POMALYST REMS™ program and be willing and able to comply with the requirements of the POMALYST REMS™ program

Exclusion Criteria:

* Patients for whom there is the prospect of stem cell transplantation in the next 6 months in the treatment plan are excluded
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia
* Waldenström's macroglobulinemia or immunoglobulin M (IgM) myeloma
* Radiotherapy to multiple sites or immunotherapy within 4 weeks before start of protocol treatment (localized radiotherapy to a single site at least 1 week before start is permissible)
* Participation in an investigational therapeutic study within 3 weeks or within 5 drug half lives (t1/2) prior to first dose, whichever time is greater
* Patients known to be refractory to any proteasome inhibitor other than bortezomib or carfilzomib
* Pregnant or lactating
* History of allergy to mannitol or prior hypersensitivity to thalidomide, lenalidomide or pomalidomide
* Major surgery within 3 weeks prior to first dose,
* Prior peripheral stem cell transplant within 12 weeks of study enrollment
* Has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal (with the exception of hormones for thyroid conditions or estrogen replacement therapy [ERT]), or any investigational therapy within 21 days of enrollment
* Myocardial infarction within 6 months prior to enrollment, New York Heart Associate (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Uncontrolled hypertension or diabetes
* Acute active infection requiring systemic antibiotics, antivirals, or anti fungals within two weeks prior to first dose
* Known or suspected human immunodeficiency (HIV) infection, known HIV seropositivity
* Active hepatitis A, B, or C infection
* Non-hematologic malignancy within the past 3 years except adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix or breast, prostate cancer < Gleason grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
* Any clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Significant neuropathy (grades 3-4, or grade 2 with pain) at the time of the first dose and/or within 14 days before enrollment
* Contraindications to any of the required concomitant drugs, including proton-pump inhibitor (eg, lansoprazole), enteric-coated aspirin, allopurinol or if a history of prior thrombotic disease, warfarin or low molecular weight heparin
* Subjects in whom the required program of PO and IV fluid hydration is contraindicated, eg, due to pre-existing pulmonary, cardiac, or renal impairment
* Subjects with known or suspected amyloidosis of any organ
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis
* Prior exposure to daratumumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08-13 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of carfilzomib when administered in combination with pomalidomide and dexamethasone | 28 days
Partial response rate after 4 courses according to International Myeloma Working Group (IMWG) criteria | 4 months
  The proportion and exact 95% binomial confidence interval for the response rate will be reported adjusted for the two-stage design of this trial.
Response rates of carfilzomib, pomalidomide, dexamethasone, and daratumumab dosing according to International Myeloma Working Group (IMWG) criteria | 4 months

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years
  Defined as at least a partial response to therapy, will be reported along with its exact 95% binomial confidence
Time to progression | Up to 2 years
  Estimated using the product-limit method of Kaplan and Meier.
Duration of response | From the date of the clinical examination which confirmed the response, until the date of disease progression, or censoring at the date of last clinical follow-up up to 2 years
  Assessed conditional upon achieving at least a partial response.
Progression-free survival | From the date of first therapy until the date of documented disease progression or death up to 2 years
  Estimated using the product-limit method of Kaplan and Meier.
Overall survival | Up to 2 years
  Estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (5):
- United States (4):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University - Karmonos Cancer Center, Detroit, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
- University Health Network - Princess Margaret Cancer Center, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Derman BA, Zonder J, Reece D, Cole C, Berdeja J, Stefka AT, Major A, Kin A, Griffith K, Jasielec J, Jakubowiak AJ. Phase 1/2 study of carfilzomib, pomalidomide, and dexamethasone with and without daratumumab in relapsed multiple myeloma. Blood Adv. 2023 Oct 10;7(19):5703-5712. doi: 10.1182/bloodadvances.2022008866. PMID 36763537